CLINICAL TRIAL: NCT02145819
Title: Optimal Planning of a Day 3 Cryopreserved(Frozen)-Thawed Embryo Transfer in a Natural Cycle With hCG Administration or After Spontaneous LH Peak?
Acronym: PLUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Arne van de Vijver, Medical Doctor, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Single Group | Purpose: Treatment
Other Study IDs: PLUS
Record Dates: First submitted 2014-01-08; First posted 2014-05-23 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Supervision of Pregnancy Resulting From In-vitro Fertilization

ARMS (2):
- A: spontaneous LH peak (Placebo Comparator): In group A, embryos are thawed 4 days after LH surge, with a re-evaluation and transfer 5 days after LH surge.
  Interventions: Other: LH peak
- B: hCG (Active Comparator): In group B, embryos are thawed 5 days after hCG administration, with a re-evaluation and transfer 6 days after hCG.
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: hCG
  Other Names: spontaneous LH peak
  Arms: B: hCG
Other: LH peak
  Arms: A: spontaneous LH peak

SUMMARY:
The aim of the study is to determine whether spontaneous LH peak is superior to human chorionic gonadotropin before a transfer of a day 3 frozen embryo.

DETAILED DESCRIPTION:
For surplus embryos after fresh IVF-cycles, cryopreservation has become common medical practice. These frozen embryos are mostly replaced in an artificial cycle with exogenous estrogen and progesterone or in a natural cycle. Often, hCG is administered as an ovulation induction agent for scheduling purposes.

Successful implantation requires a co-ordinated series of events allowing a timely dialogue between a receptive endometrium and the intrusive blastocyst . The period of receptivity is thought to be 3 days in human. It is suggested that blastocyst apposition begins about day LH+6 and is completed by day LH+10

In general, the aim is to transfer the embryo during the 'window of implantation', what is defined as the period during which the uterus is receptive for implantation of the free-lying blastocyst. This has been a subject of debate since many years.

A prospective study by Fatemi et al. (2010) revealed a significantly higher ongoing pregnancy rate after transferring frozen-thawed embryos in natural cycles with a spontaneous LH peak compared with natural cycles controlled by hCG for final oocyte maturation and ovulation (31.1% vs. 14.3%, respectively). In this trial, FrET (frozen embryo transfer) was planned 5 days after the LH surge or 5 days after the administration of 5000IU of hCG.

In order to optimize the synchronization in the hCG group, and therefore enhance the pregnancy rates, the aim is to plan a FrET 6 days after hCG administration instead of 5 days. The rationale behind is that day 3 frozen embryos are thawed the day before embryo transfer, which means they are already at day 4 of the embryonic development.

ELIGIBILITY:
Inclusion Criteria:

* Natural cycles, in which a frozen-thawed day 3 embryo is replaced.
* Signed informed consent.
* Regular cycle (i.e. between 26 and 35 days)
* Normal transvaginal ultrasound at screening, without evidence of clinically significant abnormality consistent with finding adequate for ART with respect to uterus and adnexa.
* Embryos frozen by vitrification.
* Single or dual embryo transfer.

Exclusion Criteria:

* Known allergic reactions to progesterone products.
* Intake of experimental drug within 30 days prior to study start.
* Contraindication for pregnancy.
* Embryos of women above 39 years of age at the time of embryo freezing.
* Recipients of oocyte donation cycles

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2014-01; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate | 7 weeks
  We evaluate the pregnancy, at 7 weeks amenorrhoea. Outcome is clinical pregnancy rate

SECONDARY OUTCOMES:
number of monitoring visits at the clinic per cycle | 7 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Reproductive Medicine CRG, Jette, Brussels Capital, Belgium

REFERENCES:
- [Derived] Mackens S, Stubbe A, Santos-Ribeiro S, Van Landuyt L, Racca A, Roelens C, Camus M, De Vos M, van de Vijver A, Tournaye H, Blockeel C. To trigger or not to trigger ovulation in a natural cycle for frozen embryo transfer: a randomized controlled trial. Hum Reprod. 2020 May 1;35(5):1073-1081. doi: 10.1093/humrep/deaa026. PMID 32395750